CLINICAL TRIAL: NCT01391689
Title: Evaluation of Diindolylmethane Supplementation to Modulate Tamoxifen Efficacy in Breast Cancer The Diindolylmethane Efficacy Study
Brief Title: Diindolylmethane in Treating Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0366-04; NCI-2011-00710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA149417-01A1 (NIH)
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-04

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (antineoplastic therapy) (Experimental): Patients receive diindolylmethane (BioResponse) PO BID for approximately 18 months.
  Interventions: Dietary Supplement: diindolylmethane
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for approximately 18 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: diindolylmethane — Given PO
  Other Names: DIM
  Arms: Arm I (antineoplastic therapy)
Dietary Supplement: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This phase II/III trial studies how well diindolylmethane (DIM) works and compares it to placebo in treating patients with breast cancer. DIM may slow the growth of tumor cells and be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess change in breast density using mammogram-based breast density measures as well as a novel, quantitative fat-water ratio breast magnetic resonance imaging (FWR-MRI).

II. Evaluate the effect of an escalating daily dose of DIM on serum steroid hormones (estrogen, sex hormone binding globulin [SHBG]) and urinary 2-hydroxyestrone:16 alpha-hydroxyestrone (2OHE1:16 alpha OHE1) ratio as well as serum tamoxifen (TAM) metabolites (endoxifen). The study will be initiated at a dose of 75 mg twice daily (BID) (total daily dose of 150 mg) for the first 10 study participants and then the dose will be escalated to 150 mg DIM BID (total daily dose of 300 mg) if no treatment-related serious adverse events (SAEs) are reported in the initial 10 subjects thru 3 months of treatment.

III. Expand on currently available toxicity and safety of DIM-TAM combination by assessing reports of treatment associated side effects/adverse events including TAM-associated endometrial toxicity (self-reported vaginal bleeding patterns and physician ordered vaginal ultrasound), chemistry profiles, Functional Assessment of Cancer Therapy-Endocrine Subscale (FACT-ES) scores and standard Common Terminology Criteria for Adverse Events (CTCAE) tracking.

SECONDARY OBJECTIVES:

I. Collect fine-needle aspiration breast tissue samples (in a subset) and blood samples (all participants) in order to explore change in mammary gland tissue architecture and cellularity; and tissue markers and their association with change in breast density and to explore changes in biomarkers of disease risk (e.g. cyclooxygenase-2 [COX-2], deoxyribonucleic acid [DNA] adducts, oxidative stress, inflammation, etc) over time (pre and post treatment) in both study arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive diindolylmethane orally (PO) BID for approximately 36 months.

ARM II: Patients receive placebo PO BID for approximately 36 months.

In both arms, treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed TAM as adjuvant therapy for early stage (0, I, II, IIIa) breast cancer or as chemoprevention in women at high risk for breast cancer
* New or planned prescription of TAM therapy; ineligible for randomization until on TAM for > 3 months with the expectation to continue use for > 18 months
* Mammogram with Breast Imaging Reporting and Data System (BIRADS) score of >= 2; (equivalent to the following and similar breast density descriptive terms found in mammogram reports: 2 = scattered fibroglandular elements/densities; 3 = heterogeneously dense tissue; 4 = extremely dense tissue)
* No use of soy-based dietary supplements or willingness to discontinue use, complete a 4-week wash-out period, prior to randomization, and refrain from use during trial period
* If pre-menopausal, non-pregnant (confirmed with urinary pregnancy test); practicing birth control or s/p oophorectomy
* Able to complete study run-in activities, including taking study-provided placebo pill twice daily (AM & PM) and recording pill intake and any symptoms experienced on a study calendar, with a compliance rate of at least 80%
* Normal blood chemistry test that includes sodium and specific kidney and liver function tests (creatinine, alanine amino transferase-ALT, aspartate amino transferase-AST) within 30 days of study enrollment; (Informed Consent Form signed)
* No history of hyponatremia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Urinary 2OHE1:16alpha OHE1 ratio | Up to 18 months
  estrogen metabolites measured in ng/100ul; this outcome will also be reported as a ratio

SECONDARY OUTCOMES:
Plasma TAM metabolites (ng/mL) | Up to 18 months
  measures of 4 primary metabolites (UCSF)
Serum Estrogen (estradiol) (pg/mL) | Up to 18 months
  measured at U Michigan
Self reported vaginal bleeding | Up to 24 months
  If vaginal ultrasound is available via medical records, toxicity will be addressed through endometrial evaluation. Otherwise, evaluation will be based on self report.
mammographic density | up to 18 months
  assessed by fat:water ratio magnetic resonance imaging AND mammographic density from clinical mammograms

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Thomson, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Thomson CA, Chow HHS, Wertheim BC, Roe DJ, Stopeck A, Maskarinec G, Altbach M, Chalasani P, Huang C, Strom MB, Galons JP, Thompson PA. A randomized, placebo-controlled trial of diindolylmethane for breast cancer biomarker modulation in patients taking tamoxifen. Breast Cancer Res Treat. 2017 Aug;165(1):97-107. doi: 10.1007/s10549-017-4292-7. Epub 2017 May 30. PMID 28560655